CLINICAL TRIAL: NCT07386431
Title: The Association Between Deep Endometriosis and the Occurrence of Colorectal Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Other Study IDs: 20250256
Record Dates: First submitted 2026-01-26; First posted 2026-02-04 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-06

CONDITIONS: Endometriosis; Deep Endometriosis; Bowel Endometriosis; Colorectal Carcinoma; Colon Resection; Endometriosis Pelvic; Endometriosis Rectum; Carcinogenesis; Genetic Change; Infertility
MeSH Terms: conditions — Endometriosis; Colorectal Neoplasms; Carcinogenesis; Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Biopsy of the bowel with endometriotic nodule and healthy part of bowel
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to identify the molecular or genetic mechanisms that may predispose patients with bowel endometriosis to an increased risk of colorectal carcinoma. The study will include patients for whom surgical treatment of bowel endometriosis is clinically indicated.

This research would represent a significant advancement in evaluating the necessity of surgical intervention in asymptomatic patients or those with mild symptoms. Furthermore, it would provide a broader insight into the systemic impact of endometriosis on other organ systems, ultimately improving risk assessment and preventive measures.

ELIGIBILITY:
Inclusion Criteria:

Female patients aged 18 and over, treated at the Department of Reproduction for diagnosed deep endometriosis, including bowel endometriosis, for whom surgical treatment is indicated.

Exclusion Criteria:

* Patients with known inflammatory bowel disease (IBD), patients with a personal history of gynecological or gastrointestinal malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Endometriosis is a disease that most commonly affects women.
Study Population: Female patients aged 18 and over, treated at the Department of Reproduction for diagnosed deep endometriosis, including bowel endometriosis, for whom surgical treatment is indicated.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Comparison of gene expression in healthy and with endometriosis affected bowel. | 3 years

IPD SHARING:
Plan to Share IPD: No